CLINICAL TRIAL: NCT06909955
Title: The Effect of Progressive Muscle Relaxation Exercises on Premenstrual Syndrome, Anxiety, and Tendency to Violence in Young Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mehtap kilicoz, physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7751
Record Dates: First submitted 2025-02-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Premenstrual Disorder
Keywords: premenstrual syndrome; progressive relaxation exercise
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Other: Exercise
- Control group (No Intervention)

INTERVENTIONS:
Other: Exercise — Relaxation Exercises (Progressive Muscle Relaxation Exercises):
  Progressive muscle relaxation exercises, one of the relaxation techniques, will be used in this study. Participants will be instructed to sit in a comfortable position on a chair during the exercises. Clear and precise instructions will be provided to ensure proper execution. The exercise program will be conducted for 8 weeks, 3 days a week, for 30 minutes, under the supervision of an expert physiotherapist.
  Arms: Exercise group

SUMMARY:
This study results will provide evidence on the effectiveness of Progressive Muscle Relaxation Exercises (PMRE) as a complementary method in improving Premenstrual Syndrome (PMS), an important women's health issue. Additionally, it will contribute to the literature by shedding light on irritability and anxiety, which are common side effects of PMS.

ELIGIBILITY:
Inclusion Criteria:

* Female students studying at Istanbul Aydın University, Faculty of Health Sciences, Those who score 111 or above on the Premenstrual Syndrome Scale (PMSS), Female students aged 18-24 will be included in the study.

Exclusion Criteria:

* Non-Turkish speakers, Individuals who cannot communicate normally, Students who are unable to comply with the exercise program will be excluded from the study.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only femle persons will accept
Enrollment: 84 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | evaluations will be conducted at the day 1 and after 8 weeks.
  Premenstrual Syndrome Scale (PMSS):
  Developed by Gençdoğan in 2006, this scale consists of 44 items in a five-point Likert format, with response options scored from 1 to 5.
Violence Tendency Scale | evaluations will be conducted at the day 1 and after 8 weeks.
  Violence Tendency Scale (VTS):
  Developed by Göka, Bayat, and Türkçapar (1995) for the Ministry of National Education to assess violence tendencies in secondary school students, the scale was later redesigned and validated in the Prime Ministry Family Research Institution's 1998 study on violence in family and society.
Beck Anxiety Inventory | evaluations will be conducted at the day 1 and after 8 weeks.
  Beck Anxiety Inventory (BAI):
  Developed by Beck and colleagues in 1988, the Beck Anxiety Inventory (BAI) consists of 21 items and follows a Likert-type (0-3) self-report format (Beck, Brown, Epstein, & Steer, 1988).

IPD SHARING:
Plan to Share IPD: No